CLINICAL TRIAL: NCT06584578
Title: Effect of 12 Weeks of Different Exercise Training Modalities and Nutritional Guidance on Body Composition
Brief Title: Exercise Nutrition and Body Composition
Acronym: FitNutrBC-12
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Neslihan AKÇAY, Assoc. Prof. Dr., Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKarabuk-1
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Overweight; Weight Loss; Muscle Maintenance
Keywords: Exercise; WB-EMS; Pilates; Yoga; Nutritional Guidance; Body Composition
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity | interventions — Exercise Movement Techniques; Aquatic Therapy; Tai Ji; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were strictly separated and think their intervention is the main intervention. The same is true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Whole-Body Electomyostimulation (WB-EMS) (Experimental): Whole-Body Electromyostimulation
  Interventions: Other: Whole-Body Electromyostimulation
- Pilates (Experimental): Pilates
  Interventions: Other: Pilates
- Tai Chi (Experimental): Tai-Chi exercise
  Interventions: Other: Tai Chi
- Nutrition counseling (Active Comparator): Nutrition counseling for 12 weeks
  Interventions: Other: Nutritional counseling

INTERVENTIONS:
Other: Whole-Body Electromyostimulation — Participants were included in tree exercise programs (Yoga, Pilates, WB-EMS) by an expert trainer 2 days a week for 12 weeks. At the same time, an active control group conducted a weekly diet counseling for 12 weeks by an expert dietician.
  Other Names: Whole-Body Electromyostimulation exercise; Pilates exercise; Tai Chi exercise
  Arms: Whole-Body Electomyostimulation (WB-EMS)
Other: Pilates — Pilates exercise twice weekly for 12 weeks
  Arms: Pilates
Other: Tai Chi — Pilates exercise twice weekly for 12 weeks
  Arms: Tai Chi
Other: Nutritional counseling — Nutritional counseling for 12 weeks
  Arms: Nutrition counseling

SUMMARY:
Effect of 12 Weeks of Different Exercise Training Modalities and Nutritional Guidance on Body Composition

The purpose of the study was to examine the effect of 12 weeks of different exercise training modalities and nutritional guidance on body composition.This study was conducted voluntarily by individuals who applied to a private health center in the Safranbolu district of Karabük and received medical nutrition treatment. It was conducted on four groups as Pilates, Yoga, WB-EMS and control and lasted 12 weeks in total. The training period of the participants in the group other than the control group was 2 days a week and 45 minutes per day, and 3 exercises consisted of warm-up, main part and cool-down parts. Some body composition assessments were made to the participants before and after their 12-week exercises. Body composition measurements (height, body weight, body mass index, body fat and muscle percentage) and systolic and diastolic blood pressure measurements were taken. Maximum heart rate (HRmax) (beats/min), average HR (beats/min), total calories burned (kcal) were determined to determine and monitor the load and intensity of each exercise for 12 weeks, and the Borg Scale was applied to the participants after each exercise to determine the degree of difficulty they perceived from the exercise they did and to evaluate their enjoyment of the exercises. Also, A personalized nutrition program prepared by a specialist dietitian for 12 weeks.

DETAILED DESCRIPTION:
Height and Body Composition Measurements: Height measurements of the athletes participating in the study were made with a height scale with a precision of 0.01 mm. Body weight and body mass index measurements were determined with an INBODY 120 brand body fat analyzer.

Warm-up Protocol: participants performed the same warm-up protocol in all conditions, a general warm-up consisting of 10 min of full-body light stretching exercises (do Carmo et al. 2021).

Determination of Exercise Load and Intensity: In order to determine and follow the load and intensity of each exercise for 6 weeks, a Realtrack Seego brand pulse monitoring system (Spain) was used, which instantly records the maximum heart rate (HRmax) (beats/min), average HR (beats/min), and total calories burned (kcal) values, and the values were recorded by the researcher by watching them on the monitor.

Yoga Exercise Program: Each yoga session lasts 1.5 hours. The emphasis in yoga classes is on asana practice; all types of poses are included, including sitting, standing, balancing poses, kneeling, forward and backward bending, supine and prone positions and inversions. Classes always begin with a short body and breath scan and end with an 8-10 minute relaxation practice in Savasana (lying corpse pose). The scenarios for the sessions are prepared according to two valuable yoga books (Satyananda, 2002). Yoga trainings are performed by an expert trainer.

Pilates Exercise Program: The Pilates exercise program complied with the recommended amount of exercise for improving the health of the elderly, and the movements suitable for the elderly were selected from the work of Cathleen Murakami (Murakami, 2006). The Pilates exercise program included a five-minute warm-up exercise, and the order was as follows: breathing, 2 repetitions (repetitions); compression and release, 2 repetitions × 2 sets; supine spine, 2 repetitions × 2 sets; arm circles, 4 repetitions × 2 sets; knee-to-knee bending stretch, 2 repetitions × 2 sets; pelvic peel and hinge, 2 repetitions × 2 sets; arms crossed spine, 2 repetitions × 2 sets; and seated hip stretch, 2 repetitions. The main exercise was performed for 30 minutes in the following order: swim, 10 repetitions × 1 set; rolling and rolling, 3 repetitions × 2 sets; single leg circle, 5 repetitions × 2 sets. The cool-down exercise was performed in the same way as the warm-up exercise (Herman, 2008). Pilates training was performed by an expert trainer.

Nutritional Guidance: A personalized nutrition program was prepared for each participant by a dietician in a face-to-face meeting based on the individual's body analysis values (body fat, muscle mass, body water ratios), complete blood count results, lifestyle and eating habits, with daily calorie intake not below the Basal Metabolic Rate (BMR) and a protein value of at least 1.5 g/kg.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Willing to maintain the intervention for 12 weeks

Exclusion Criteria:

* Being under 18 years old
* Having a chronic disease
* Medication that relevantly affect muscle metabolism
* Contraindication for Bio Impedance Analysis
* Contraindication for Whole Body Electromyostimulation
* Contraindications for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Muscle mass changes from baseline assessment to 12 week follow-up assessment | From baseline assessment to 12 week follow-up assessment
  Muscle mass changes from baseline assessment to 12 week follow-up assessment as determined my Bio Impedance Analysis

SECONDARY OUTCOMES:
Body Fat Content changes from baseline assessment to 12 week follow-up | From baseline assessment to 12 week follow-up assessment
  Changes of Body Fat Content (in %) from baseline assessment to 12 week follow-up assessment as determine by Bio Impedance Analysis
Body Fat Mass changes from baseline assessment to 12 week follow-up assessment | From baseline assessment to 12 week follow up assessment
  Body Fat Mass (kg) changes from baseline assessment to 12 week follow up assessment as determine by Bio Impedance Analysis
Body mass changes from baseline assessment to 12 week follow-up assessment | From baseline assessment to 12 week follow-up assessment
  Changes of body mass (weight in kg) from baseline assessment to 12 week follow-up assessment as determined by Bio Impedance Analysis
Body water changes from baseline assessment to 12 week follow-up assessment | From baseline assessment to 12 week follow-up assessment
  Changes of body water from baseline assessment to 12 week follow-up assessment as determined by Bio Impedance Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan AKÇAY, Doctorate, Study Chair — Karabuk University
Locations (1):
- Karabuk University, Karabük, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Willert S, Weissenfels A, Kohl M, von Stengel S, Frohlich M, Kleinoder H, Schone D, Teschler M, Kemmler W. Effects of Whole-Body Electromyostimulation on the Energy-Restriction-Induced Reduction of Muscle Mass During Intended Weight Loss. Front Physiol. 2019 Aug 12;10:1012. doi: 10.3389/fphys.2019.01012. eCollection 2019. PMID 31456693
- [Background] Kemmler W, Weissenfels A, Teschler M, Willert S, Bebenek M, Shojaa M, Kohl M, Freiberger E, Sieber C, von Stengel S. Whole-body electromyostimulation and protein supplementation favorably affect sarcopenic obesity in community-dwelling older men at risk: the randomized controlled FranSO study. Clin Interv Aging. 2017 Sep 21;12:1503-1513. doi: 10.2147/CIA.S137987. eCollection 2017. PMID 28989278